CLINICAL TRIAL: NCT02895633
Title: Osteoarticular Tumor Characterization by Advanced Imaging
Acronym: TUMOSTEO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009-A00758-49
Record Dates: First submitted 2016-09-05; First posted 2016-09-12 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Bone Tumor; Soft Tissue Tumor
Keywords: MR imaging; Diffusion weighted imaging; MR proton spectroscopy; CT perfusion; Contrast enhanced ultrasound
MeSH Terms: conditions — Bone Neoplasms; Soft Tissue Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with bone or peripheral soft-tissue tumor (Experimental)
  Interventions: Other: Ecography; Other: CT scan; Other: MRI

INTERVENTIONS:
Other: Ecography — Standard Doppler ultrasound and perfusion imaging after injection of Sonovue
Other: CT scan — With injection of Iomeron 400
Other: MRI — With injection of gadolinium (Multihance)

SUMMARY:
The purpose is to compare and evaluate multiple functional imaging methods (perfusion, diffusion, spectroscopy) for initial benign/malignant characterization of osteoarticular tumors and to determine which method or which association of methods could improve non invasive tissue characterization.

Secondary purposes are:

* to determine a possible correlation between some parameters and the histological grade (FNCLCC)
* to suggest a coherent diagnostic imaging approach for osteoarticular tumors.

The ancillary study will enroll patients needing radiological tumor follow-up. The purpose is to identify tools for evaluation of tumor activity and therapeutic response before modification of morpho-volumetric data.

DETAILED DESCRIPTION:
Patients refered for the initial evaluation of suspected osteoarticular masses will be included in this study after signing an informed consent.

Histologic analysis will be used as a gold standard.

The following imaging techniques will be evaluated:

* contrast enhanced ultrasonography
* Low dose CT perfusion
* Magnetic resonance perfusion
* Diffusion weighted imaging
* Magnetic resonance proton spectroscopy

ELIGIBILITY:
Inclusion Criteria:

* patients examined for initial assessment of bone or peripheral soft-tissue primitive tumor
* patients with normal awareness level
* patients having signed informed consent

Exclusion Criteria:

* pregnant women
* persons deprived of liberty
* persons under legal protection or unable to give informed consent
* persons in life-threatening emergency
* allergy to Sonovue, iodinated contrast media or gadolinium chelates
* risk of pregnancy
* breastfeeding women
* acute coronary syndrome or unstable ischemic cardiopathy (ban on injection of contrast agent for CT scan)
* renal failure (ban on injection of contrast agent for MRI and CT scan)
* contraindication to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1090 (Estimated)
Dates: Start 2009-11; Primary Completion 2018-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Contrast enhancement in echography: yes or no | baseline
Contrast enhancement curve (absent, slow or fast) in echography | baseline
Maximal intensity of enhancement peak in echography | baseline
Mean transit time of enhancement in echography | baseline
Gradient of contrast enhancement curve in echography | baseline
Vascularization (dynamic analysis) in CT scanner | baseline
  * 0: absent
  * 1: low (< 20UH)
  * 2: > 20 UH without new blood vessels
  * 3: > 20 UH and/or with new blood vessels
Contrast enhancement curve (absent, slow or fast) in CT scanner | baseline
Maximal intensity of enhancement peak in CT scanner | baseline
Mean transit time of enhancement in CT scanner | baseline
Gradient of contrast enhancement curve in CT scanner | baseline
Contrast enhancement curve (absent, slow or fast) in MRI | baseline
Maximal intensity of enhancement peak in MRI | baseline
Mean transit time of enhancement in MRI | baseline
Gradient of contrast enhancement curve in MRI | baseline
Choline peak in magnetic resonance spectroscopy | baseline
  Choline presence was defined as a clear metabolite peak at 3.2 ppm
Apparent diffusion coefficient (ADC) in MR diffusion weighted imaging | baseline
  ADC value in mm2/s
Area under the perfusion curve in MRI | baseline
Perfusion curve gradient in MRI | baseline
Perfusion time-to-peak in MRI | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Augusto GONDIM TEIXEIRA, Principal Investigator — Service d'Imagerie Guilloz, CHRU Nancy
Locations (1):
- Service d'Imagerie Guilloz, CHRU Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ribeiro GJ, Gillet R, Hossu G, Trinh JM, Euxibie E, Sirveaux F, Blum A, Teixeira PAG. Solitary bone tumor imaging reporting and data system (BTI-RADS): initial assessment of a systematic imaging evaluation and comprehensive reporting method. Eur Radiol. 2021 Oct;31(10):7637-7652. doi: 10.1007/s00330-021-07745-9. Epub 2021 Mar 25. PMID 33765161